CLINICAL TRIAL: NCT05416463
Title: A Single-blinded Randomized Control Study and Economic Analysis of an Intraoperative Navigation System for Total Hip Arthroplasty
Brief Title: Clinical Study and Economic Analysis of an Intraoperative Navigation System for Total Hip Arthroplasty
Acronym: INSTHA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Grand River Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INSTHA
Record Dates: First submitted 2022-06-07; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Total Hip Arthroplasty
MeSH Terms: interventions — Tacrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Sham Comparator): The control group will receive primary elective THA as per standard of care surgical protocols for this type of surgery
  Interventions: Procedure: Intra-Operative Device for THA
- Treatment (Experimental): The intervention group will receive primary elective THA with the use of Intellijoint HIP 3D mini-optical navigation tool.
  Interventions: Procedure: Intra-Operative Device for THA

INTERVENTIONS:
Procedure: Intra-Operative Device for THA — The intervention group will receive primary elective THA with the use of Intellijoint HIP 3D mini-optical navigation tool.

SUMMARY:
This study will assess the clinical and health economic value of an intraoperative navigation system for total hip arthroplasty in one Ontario hospital. The results of this study will be used to generate evidence-based recommendations on the use and funding of the device in public hospitals and inform the development of a provincial healthcare innovation pathway.

ELIGIBILITY:
Inclusion Criteria:

* Receiving primary THA
* Elective THA
* Provision of informed consent

Exclusion Criteria:

* Unable to obtain informed consent
* Receiving revision THA
* THA is to treat trauma (i.e. hip fracture and/or dislocation)
* Patient is undergoing simultaneous bilateral hip replacement
* Performing surgeon is not participating in the study
* Hip fracture
* Hip dislocation
* Severe osteoporosis
* Trochanteric osteotomy
* Suspected or actual infection
* Existing implanted hardware
* Severe deformities of the femoral or pelvic bone
* High Body Mass Index (BMI)*

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Activities of Daily Living | up to 12 months
  Hip disability and Osteoarthritis Outcome Score (HOOS)
  Scores are 1-100 and each subscale is scored and then connected with a line on a graph to generate a "HOOS profile".
  "0 indicates extreme problems and 100 indicates no problems."

IPD SHARING:
Plan to Share IPD: No